CLINICAL TRIAL: NCT02891135
Title: Randomized Evaluation of a Simplified Clinical Algorithm for Identifying Patients Eligible for Immediate Initiation of Antiretroviral Therapy for HIV
Brief Title: Simplified Algorithm for Treatment Eligibility
Acronym: SLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Sydney Rosen, Principal Investigator, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-35634
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: HIV
Keywords: WHO 'Treat all" Antiretroviral Guidelines; Simplified Algorithm for Treatment Eligibility (SLATE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Patients randomized to the standard arm will receive standard procedures for initiating antiretroviral therapy for HIV.
- Intervention (Experimental): Patients randomized to the intervention arm will be offered immediate treatment initiation under the intervention algorithm (SLATE).
  Interventions: Other: SLATE

INTERVENTIONS:
Other: SLATE — Algorithm for collecting information required to determine if patient is eligible for immediate (same-day/same-visit) initiation of antiretroviral medications.
  Arms: Intervention

SUMMARY:
In its 2015 revision of the global guidelines for HIV care and treatment, the World Health Organization called for initiating lifelong antiretroviral treatment (ART) for all patients testing positive for HIV, regardless of CD4 cell count. As countries adopt the new recommendation, known as "treat all," millions of additional patients are becoming eligible for ART worldwide. In sub-Saharan Africa, where most of these patients are located, studies continue to document high losses of treatment-eligible patients from care before they receive their first dose of antiretroviral medications. Among facility-level reasons for these losses are treatment initiation protocols that require multiple clinic visits and long waiting times before a patient who tests positive for HIV is dispensed an initial supply of medications. Simpler, more efficient, accelerated algorithms for ART initiation will be needed if "treat all" is to realize the benefits expected.

Experts have proposed a simplified clinical algorithm to screen patients for eligibility for immediate ART initiation at a patient's first clinic visit, without the use of point-of-care laboratory test technologies. The Simplified Algorithm for Treatment Eligibility (SLATE) uses four screens to assess whether a patient is eligible for same-day treatment initiation: i) symptom report, ii) medical history, iii) brief physical examination; and iv) readiness assessment. SLATE is a pragmatic, individually randomized evaluation to determine the effectiveness of the algorithm in increasing ART initiation among non-pregnant adult patients. Approximately 960 HIV-infected adult patients not yet on ART will be enrolled during a routine clinic visit and randomized to receive the intervention or standard care. Patients in the intervention arm will be administered the SLATE screens; those found eligible under the algorithm will be offered immediate treatment initiation, while those who are not eligible will be referred for standard clinic care. Patients in the standard arm will be referred for ART initiation under standard clinic procedures. All care after the initial visit will be by the clinic under standard of care. If successful, SLATE will offer a standardized approach to collecting and interpreting a minimum set of patient data that will avoid delaying treatment initiation for the majority of patients who are eligible for immediate ART, while deferring initiation in the minority who should not start immediately.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) (initiating children on ART is likely to require additional information, making the SLATE algorithm less applicable to pediatric populations)
* Confirmed HIV-positive test result at any time (may have been diagnosed previously)
* Not currently on ART (three-drug combination)
* Presented at the study clinic for any HIV-related reason, including an HIV test, pre-ART monitoring, or ART initiation

Exclusion Criteria:

* Pregnant (pregnancy is an exclusion criterion because treatment guidelines for pregnant women differ from those for non-pregnant adults; most pregnant women are diagnosed with HIV and initiated on ART in antenatal clinics, not general adult HIV clinics)
* Not intending to return to this clinic for further HIV care in the coming year (i.e. intends to seek further care somewhere else)
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff
* Not willing or able to provide written informed consent to participate in the study
* Previously enrolled in the same study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment initiation | 28 days after study enrollment
  Proportion of patients initiated on ART within 28 days of study enrollment
Treatment initiation and retention | 8 months after study enrollment
  Proportion of patients who initiate ART within 28 days of study enrollment and are alive, in care, and retained on ART eight months after study enrollment

SECONDARY OUTCOMES:
Initiation within 14 days | 14 days after study enrollment
  Proportion of patients who initiate ART within 14 days of study enrollment
Viral suppression | 8 months after study enrollment
  Proportion of patients who are virally suppressed according to local guidelines within 8 months of study enrollment
One-year retention in care | 14 months after study enrollment
  Retention defined as > 1 month late for last scheduled visit
One-year retention in care | 16 months after study enrollment
  Retention defined as > 3 months late for last scheduled visit
SLATE eligibility | Study enrollment
  Proportions of HIV-positive patients presenting at study clinics and not yet on ART who are eligible and ineligible for immediate initiation using SLATE algorithm criteria
SLATE ineligibility reasons | Study enrollment
  Reasons for ineligibility for immediate initiation, among those found ineligible in the intervention arm
Time to initiation | 8 months
  Average time to ART initiation (days) for each arm

OTHER OUTCOMES:
Patient preferences | Study enrollment
  Patient preferences on the speed and timing of ART initiation
Patient costs | 8 months
  Costs to patients of ART initiation under standard and intervention procedures
Provider costs | 8 months
  Costs to providers of ART initiation under standard and intervention procedures

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, Principal Investigator — Boston University
Locations (2):
- Kenya Medical Research Institute/Walter Reed Projects, Kericho, Kericho County, Kenya
- Health Economics and Epidemiology Research Office, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be retained in secure study databases until completion of the study, including completion of all data analysis and report writing associated with the study and closing of the IRB-approved protocol. Study data sets and other electronic files containing study data will then have all identifiers removed and where possible will be made available for use of other researchers through a repository such as Dryad.

REFERENCES:
- [Background] Rosen S, Fox MP, Larson BA, Sow PS, Ehrenkranz PD, Venter F, Manabe YC, Kaplan J; Models for Accelerating Treatment Initiation (MATI) Technical Consultation. Accelerating the Uptake and Timing of Antiretroviral Therapy Initiation in Sub-Saharan Africa: An Operations Research Agenda. PLoS Med. 2016 Aug 9;13(8):e1002106. doi: 10.1371/journal.pmed.1002106. eCollection 2016 Aug. PMID 27505444
- [Background] Fox MP, Rosen S. A new cascade of HIV care for the era of "treat all". PLoS Med. 2017 Apr 11;14(4):e1002268. doi: 10.1371/journal.pmed.1002268. eCollection 2017 Apr. PMID 28399160
- [Background] Rosen S, Fox MP, Larson BA, Brennan AT, Maskew M, Tsikhutsu I, Bii M, Ehrenkranz PD, Venter WF. Simplified clinical algorithm for identifying patients eligible for immediate initiation of antiretroviral therapy for HIV (SLATE): protocol for a randomised evaluation. BMJ Open. 2017 May 28;7(5):e016340. doi: 10.1136/bmjopen-2017-016340. PMID 28554939
- [Result] Rosen S, Maskew M, Larson BA, Brennan AT, Tsikhutsu I, Fox MP, Vezi L, Bii M, Venter WDF. Simplified clinical algorithm for identifying patients eligible for same-day HIV treatment initiation (SLATE): Results from an individually randomized trial in South Africa and Kenya. PLoS Med. 2019 Sep 16;16(9):e1002912. doi: 10.1371/journal.pmed.1002912. eCollection 2019 Sep. PMID 31525187
- [Result] Brennan AT, Maskew M, Larson BA, Tsikhutsu I, Bii M, Vezi L, Fox MP, Venter WD, Ehrenkranz P, Rosen S. Who is seeking antiretroviral treatment for HIV now? Characteristics of patients presenting in Kenya and South Africa in 2017-2018. J Int AIDS Soc. 2019 Sep;22(9):e25358. doi: 10.1002/jia2.25358. PMID 31518058
- [Derived] Maskew M, Parrott S, De Voux L, Sharpey-Schafer K, Crompton T, Govender AC, Pisa PT, Rosen S. Triaging Clients at Risk of Disengagement from HIV Care: Application of a Predictive Model to Clinical Trial Data in South Africa. Risk Manag Healthc Policy. 2025 May 16;18:1601-1619. doi: 10.2147/RMHP.S510666. eCollection 2025. PMID 40395656
- [Derived] Maskew M, Brennan AT, Venter WDF, Fox MP, Vezi L, Rosen S. Retention in care and viral suppression after same-day ART initiation: One-year outcomes of the SLATE I and II individually randomized clinical trials in South Africa. J Int AIDS Soc. 2021 Oct;24(10):e25825. doi: 10.1002/jia2.25825. PMID 34612601
- [Derived] Brennan A, Maskew M, Larson BA, Tsikhutsu I, Bii M, Vezi L, Fox M, Venter WDF, Ehrenkranz PD, Rosen S. Prevalence of TB symptoms, diagnosis and treatment among people living with HIV (PLHIV) not on ART presenting at outpatient clinics in South Africa and Kenya: baseline results from a clinical trial. BMJ Open. 2020 Sep 6;10(9):e035794. doi: 10.1136/bmjopen-2019-035794. PMID 32895266
- See also: CROI poster with preliminary results for South Africa — http://www.croiconference.org/sessions/same-day-art-initiation-slate-trial-south-africa-preliminary-results
- See also: CROI 2019 poster and video with primary outcome results for Kenya — http://www.croiconference.org/sessions/same-day-art-initiation-slate-trial-kenya-preliminary-results